CLINICAL TRIAL: NCT05729204
Title: Washing COVID-19 Away With a Hypertonic Seawater Nasal Irrigation Solution Containing Algal and Herbal Natural Ingredients
Brief Title: Washing COVID-19 Away With a Hypertonic Seawater Nasal Irrigation Solution
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Larissa University Hospital (Other)
Responsible Party: Principal Investigator, Ioannis Pantazopoulos, Assistant Professor of Emergency Medicine, Larissa University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 13149
Record Dates: First submitted 2023-02-13; First posted 2023-02-15 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: SARS-CoV2 Infection
Keywords: Nasal irrigation; Hypertonic seawater solution; SARS-CoV2; Viral load
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypertonic seawater group (Experimental): Patients that will receive nasal irrigations with hypertonic (2.3% NaCl) seawater solution containing brown algae (Undaria pinnatifida) and blue-green algae (Spirulina platensis) as well as essential oils of Eucalyptus globulus and Mentha spicata, and Thymus vulgaris extract (Sinomarin® Plus Algae Cold & Flu Relief, Gerolymatos International SA, Krioneri, Greece)
  Interventions: Other: Hypertonic seawater solution
- control group (No Intervention): Patients that will not perform nasal irrigations

INTERVENTIONS:
Other: Hypertonic seawater solution — Nasal irrigations with hypertonic seawater solution
  Other Names: Sinomarin
  Arms: Hypertonic seawater group

SUMMARY:
Nasal irrigations are thought to reduce the amount of virus from the nasal cavity. The aim of the present study is to evaluate the effect of a hypertonic seawater solution containing algal and herbal natural ingredients (Sinomarin®) on the nasopharyngeal viral load in hospitalized patients with severe COVID-19 pneumonia. The investigators will conducted a prospective, randomized, controlled trial. Patients will be allocated in two groups, the hypertonic seawater group receiving nasal irrigations with a hypertonic seawater solution (Sinomarin®) every 4 hours during a 16-hour interval per day, for two consecutive days, and the control group (no nasal irrigations). Forty-eight hours after the baseline nasopharyngeal swab (and 8 hours after the last wash in the hypertonic seawater group), a second nasopharyngeal swab will be collected for the semiquantitative estimation of the SARS-CoV-2 viral load as determined by cycle threshold (Ct) values.

DETAILED DESCRIPTION:
Investigators will perform a prospective, randomized, controlled study in 56 patients with confirmed COVID-19 pneumonia. All patients will be treated with the standard protocol of care for COVID-19 at the Department of Infectious Diseases and will be randomized into one of two groups with the method of sequentially numbered, opaque, sealed envelopes, the hypertonic seawater group (will receive a hypertonic (2.3% NaCl) seawater solution containing brown algae (Undaria pinnatifida) and blue-green algae (Spirulina platensis) as well as essential oils of Eucalyptus globulus and Mentha spicata, and Thymus vulgaris extract (Sinomarin® Plus Algae Cold & Flu Relief, Gerolymatos International SA, Krioneri, Greece)) and the control group (no treatment). Sinomarin® is a medical device that utilizes continuous flow diffusion. The solution continues to flow as long as the nozzle is pressed, providing efficient cleansing.

At admission, a baseline nasopharyngeal swab will be collected from all patients and placed in a sterile bottle containing virus transport medium (10 ml tube with 3 ml medium, Biobase, Biodustry, Shandong, China) for SARS-CoV-2 nucleic acid detection (zero hour). Patients in the hypertonic seawater group will be given a review on the proper technique for nasal irrigation. Specifically, they will be instructed to blow their nose before irrigation, gently bend their neck forward, tilt their head to one side, and insert the nozzle into the nostril in line with the nasal septum. They will be advised to press firmly on the nozzle to squirt the solution into the nostril and then repeat the process on the other nostril. The patients will also be instructed to spit out any solution coming into their mouth and then return to an upright position to allow the solution to work for a few seconds before blowing their nose gently. After each use, they will be advised to remove the nozzle from the bottle, wash it thoroughly with warm water, and wipe it dry. Thereafter, patients will be given one bottle of 200 ml Sinomarin® and will be instructed to perform nasal irrigation to each nostril every 4 hours for a 16-hour period per day, for two consecutive days.

Forty-eight hours after the baseline nasopharyngeal swab and 8 hours after the last nasal wash, a second nasopharyngeal swab will be collected for viral load measurement. All nasopharyngeal swabs will be collected by a physician blinded to group allocation and will be collected from the same nostril for each patient.

Demographic data including age, sex, nationality, body mass index, smoking status, and date of admission will be collected at baseline. Data on comorbidities, Charlson comorbidity index, disease related symptoms, vaccination status, presenting day of illness since symptom onset, oxygenation status (PaO2/FiO2), and medication administered will also be recorded. Furthermore, outcome and potential adverse effects related to use of hypertonic seawater solution containing algal and herbal natural ingredients will be recorded. All patients will be followed until hospital discharge, ICU admission, or death. Those that will be discharged will be reexamined 14 days after hospital discharge for real-time polymerase chain reaction (RT-PCR). Manual chart review will be used to gather details of the laboratory studies, course, and outcomes.

ELIGIBILITY:
Inclusion Criteria:

* adult patients hospitalized primarily for COVID-19 pneumonia
* confirmed SARS-CoV2 infection diagnosed through RT-PCR test of nasopharyngeal samples

Exclusion Criteria:

* patients with confirmed SARS-CoV2 infection who were not primarily admitted for COVID-19 pneumonia
* patients with use of intranasal sprays for at least two weeks prior to study enrollment
* sinonasal surgery within 3 months prior to study enrollment
* patients with sinusitis
* inability to perform nasopharyngeal wash
* participation in other trials

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
SARS-CoV2 viral load | 48 hours
  SARS-CoV2 viral load in nasopharyngeal swab in hospitalized patients with COVID-19 pneumonia

SECONDARY OUTCOMES:
Need for escalation to HFNC / NIV, ICU admission | From date of randomization until hospital discharge, ICU admission or date of death from any cause, whichever came first assessed up to 3 months
  Number of participants with need for escalation to high flow nasal oxygen or non-invasive ventilation or ICU admission in patients with COVID-19 pneumonia.

CONTACTS AND LOCATIONS:
Overall Officials: Ioannis Pantazopoulos, MD, Study Director — University Hospital of Larissa
Locations (1):
- University Hospital of Larissa, Larissa, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data (IPD)
Time Frame: For one year after the end of the study
Access Criteria: Contact study director by e-mail

REFERENCES:
- [Background] Pantazopoulos I, Chalkias A, Mavrovounis G, Dimeas I, Sinis S, Miziou A, Rouka E, Poulas K, Gourgoulianis K. Nasopharyngeal Wash with Normal Saline Decreases SARS-CoV-2 Viral Load: A Randomized Pilot Controlled Trial. Can Respir J. 2022 Sep 27;2022:8794127. doi: 10.1155/2022/8794127. eCollection 2022. PMID 36247079
- [Background] Kanjanawasee D, Seresirikachorn K, Chitsuthipakorn W, Snidvongs K. Hypertonic Saline Versus Isotonic Saline Nasal Irrigation: Systematic Review and Meta-analysis. Am J Rhinol Allergy. 2018 Jul;32(4):269-279. doi: 10.1177/1945892418773566. Epub 2018 May 18. PMID 29774747
- [Background] Kwon PS, Oh H, Kwon SJ, Jin W, Zhang F, Fraser K, Hong JJ, Linhardt RJ, Dordick JS. Sulfated polysaccharides effectively inhibit SARS-CoV-2 in vitro. Cell Discov. 2020 Jul 24;6(1):50. doi: 10.1038/s41421-020-00192-8. eCollection 2020. No abstract available. PMID 32714563
- [Background] Pradhan B, Nayak R, Patra S, Bhuyan PP, Behera PK, Mandal AK, Behera C, Ki JS, Adhikary SP, MubarakAli D, Jena M. A state-of-the-art review on fucoidan as an antiviral agent to combat viral infections. Carbohydr Polym. 2022 Sep 1;291:119551. doi: 10.1016/j.carbpol.2022.119551. Epub 2022 May 2. PMID 35698330
- [Background] Huijghebaert S, Hoste L, Vanham G. Essentials in saline pharmacology for nasal or respiratory hygiene in times of COVID-19. Eur J Clin Pharmacol. 2021 Sep;77(9):1275-1293. doi: 10.1007/s00228-021-03102-3. Epub 2021 Mar 27. PMID 33772626
- [Background] Ramalingam S, Graham C, Dove J, Morrice L, Sheikh A. A pilot, open labelled, randomised controlled trial of hypertonic saline nasal irrigation and gargling for the common cold. Sci Rep. 2019 Jan 31;9(1):1015. doi: 10.1038/s41598-018-37703-3. PMID 30705369
- [Background] Slapak I, Skoupa J, Strnad P, Hornik P. Efficacy of isotonic nasal wash (seawater) in the treatment and prevention of rhinitis in children. Arch Otolaryngol Head Neck Surg. 2008 Jan;134(1):67-74. doi: 10.1001/archoto.2007.19. PMID 18209140
- [Background] Gangadi M, Georgiou S, Moschotzopoulou E, Antronikou T, Kainis E, Alevizopoulos K. Efficacy and safety of a hypertonic seawater nasal irrigation solution containing algal and herbal natural ingredients in patients with COVID-19. Eur Rev Med Pharmacol Sci. 2022 Dec;26(2 Suppl):112-123. doi: 10.26355/eurrev_202212_30495. PMID 36524919